CLINICAL TRIAL: NCT04063852
Title: Impact of Percutaneous Posterior Tibial Nerve Stimulation on Urinary and Global Quality of Life in Multiple Sclerosis Patients
Brief Title: PTNS on Urinary and Global Quality of Life in MS Patients
Acronym: PTNSinMS
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Society of Urodynamics, Female Pelvic Medicine & Urogenital Reconstruction (Other)
Responsible Party: Principal Investigator, Giulia Lane, Assistant Professor, University of Michigan
Other Study IDs: HUM00153287
Record Dates: First submitted 2019-08-19; First posted 2019-08-21 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Multiple Sclerosis; Lower Urinary Tract Symptoms; Neurogenic Bladder; Overactive Bladder; Urinary Incontinence; Urinary Urge Incontinence
MeSH Terms: conditions — Multiple Sclerosis; Lower Urinary Tract Symptoms; Urinary Bladder, Neurogenic; Urinary Bladder, Overactive; Urinary Incontinence; Urinary Incontinence, Urge

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a single-centered, prospective, longitudinal, observational cohort study of patients with MS who suffer from lower urinary tract symptoms (LUTS) and are refractory to two prior treatment modalities who have elected to pursue PTNS therapy for LUTS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Multiple Sclerosis
* Lower urinary tract symptoms (urinary frequency, urgency and/or incontinence)
* Failed prior first and second line therapy (behavioral and pharmacotherapy)
* Electing for Posterior Tibial Nerve Stimulation therapy for urinary symptoms
* Patients performing Intermittent Catheterization are Eligible

Exclusion Criteria:

* Indwelling catheters (urethral or suprapubic)
* Currently pregnant or planning pregnancy
* Unable to attend weekly office visits for PTNS
* Urodynamic findings of bladder outlet obstruction

History of:

bladder reconstruction (augmentation cystoplasty, catheterizable channel) cystectomy bladder stones pacemaker or defibrillator malignancy of bladder sacral neuromodulation intravesical injection of onabotulinum toxin within 9 months

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the urology clinic at a tertiary care referral center.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2022-11-27 (Actual); Study Completion 2022-11-27 (Actual)

PRIMARY OUTCOMES:
Urinary Frequency and/or Urinary Incontinence Episodes on 3 day voiding diary | up to 24 months.
  Change from baseline in the median number of urinary frequency and/or urinary incontinence episodes on a 3 day voiding diary at 3, 12, and 24 months

OTHER OUTCOMES:
American Urological Association (AUA) Symptom Score | up to 24 months
  Change from baseline of the total AUA Symptom Score at 3, 12, and 24 months
  7 question scale. Score Ranges 0-35. Higher scores indicate worse lower urinary tract symptoms.
  AUA Bother Subscore: Single question item that is part of the AUA symptom score, but not calculated for the overall score. range is 0-6 with 6 indicating terrible bother from urinary symptoms.
Michigan Incontinence Symptom Index | up to 24 months
  Change from baseline of the total Michigan Incontinence Symptom Index at 3, 12, and 24 months
Neurogenic Bladder Symptom Score | up to 24 months
  Change from baseline of the total Neurogenic Bladder Symptom Score at 3, 12, and 24 months
  The NBSS consists of 24 questions. The first question classifies patients by bladder management, but does not make up part of the numeric score. The remaining questions address 3 domains: incontinence, storage and voiding, and consequences. The final question is an overall quality of life question. The total score can range from 0 (no symptoms at all) to 74 (maximum symptoms). The median time to complete the NBSS is 6 minutes.
Health Status Questionnaire (SF-12), | up to 24 months
  Change in from baseline of the total Health Status Questionnaire (SF-12) at 3, 12, and 24 months
  12 item scale with ranges from 0-100. where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.
Sexual Satisfaction Scale (SSS) | up to 24 months
  Change from baseline of the total Sexual Satisfaction Scale (SSS) at 3, 12, and 24 months
  Raw scores on the 4 sexual satisfaction items (Items 2-5) are summed to create a total score. Thus, this scale can range from 4-24. Higher scores indicate greater problems with sexual satisfaction.
Bowel Control Scale (BCS) | up to 24 months
  Change from baseline of the total Bowel Control Scale (BCS) at 3, 12, and 24 months
  Raw scores on the 5 items are summed to create a Bowel Control Scale (BWCS) total score. Scores can range from 0-26, with higher scores indicating greater bowel control problems.

CONTACTS AND LOCATIONS:
Overall Officials: John Stoffel, MD, Principal Investigator — University of Michigan; Giulia Lane, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lane GI, Mao-Draayer Y, Barboglio-Romo P, Clemens JQ, Gupta P, Dunn R, Qin Y, Cameron AP, Stoffel JT. A prospective observational cohort study of posterior tibial nerve stimulation in patients with multiple sclerosis: design and methods. BMC Urol. 2020 May 27;20(1):58. doi: 10.1186/s12894-020-00629-y. PMID 32460741